CLINICAL TRIAL: NCT01200901
Title: Quetiapine in Melancholic Depression: an fMRI Study of Treatment-induced Changes in the Neurocircuitry of the Stress Response
Brief Title: Quetiapine in Melancholic Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Erik Nelson, Adjunct Associate Professor, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nelson AZ-IIT
Record Dates: First submitted 2010-09-07; First posted 2010-09-14 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Depression; Healthy
Keywords: depression; healthy
MeSH Terms: conditions — Depression | interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Melancolic depression patients (Experimental): Patients with major depression will be recruited for the 8-week clinical trial of quetiapine XR 100 - 300 mg (flexible dosing).
  Interventions: Drug: Quetiapine

INTERVENTIONS:
Drug: Quetiapine — quetiapine XR 100 - 300 mg (flexible dosing)
  Other Names: Open Label Quetiapine

SUMMARY:
In summary, the investigators propose to integrate fMRI assessments within a clinical trial of quetiapine XR in patients with melancholic depression in order to test the predictions that:

1. quetiapine XR treatment will be effective and safe for patients with major depression with melancholic features
2. successful treatment with quetiapine XR will be associated with normalization of limbic areas associated with increased salivary cortisol response to a stressful task as well as normalization on the emotional faces task differences in the melancholic group compared with healthy volunteers.
3. successful treatment with quetiapine XR will be associated with normalization of the salivary cortisol response to the stressful math task (i.e. there will be a diminished post-treatment mean AUC for cortisol secretion after the stress task compared to the pre-treatment AUC values in the patient group)

DETAILED DESCRIPTION:
Patients with major depression (N=20) will be recruited for the 8-week clinical trial of quetiapine XR 100 - 300 mg (flexible dosing). Patients who consent to participate will be referred for an initial fMRI scanning session prior to the initiation of quetiapine XR. Baseline fMRI will be obtained during the index assessment prior to initiating quetiapine XR therapy and then will be re-acquired at the final study visit at 8 weeks (the time of scheduled visits). Ten demographically matched healthy subjects will receive the same fMRI investigations on two occasions in order to provide a healthy baseline comparison to permit interpretation of the patient findings (e.g., whether initial and final fMRI measures in patients are abnormal and to control for any adaptation to the task that may normally occur).

ELIGIBILITY:
Inclusion criteria

* Provision of written informed consent
* A diagnosis of major depression with melancholic features by Diagnostic and Statistical Manual of Mental Disorders- Fourth Edition (DSM-IV)
* Females and males aged 18-65 years
* Female patients of childbearing potential must be using a reliable method of contraception and have a negative urine human chorionic gonadotropin (HCG) test at enrollment
* Able to understand and comply with the requirements of the study
* Subjects will have a Hamilton Depression Rating Scale, 28-item version (HDRS-28) score of at least 20 at the baseline visit.

Exclusion criteria

* Pregnancy or lactation
* Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others
* Known intolerance or lack of response to quetiapine fumarate, as judged by the investigator
* Use of any of the following cytochrome P450 3a4 inhibitors in the 14 days preceding enrolment including but not limited to: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine and saquinavir
* Use of any of the following cytochrome P450 inducers in the 14 days preceding enrolment including, but not limited to: phenytoin, carbamazepine, barbiturates, rifampin, and St. John's Wort.
* Administration of a depot antipsychotic injection within one dosing interval (for the depot) before randomisation Women using oral contraceptives or other medications that directly affect estrogen or progesterone system in the body.
* Subjects taking corticosteroids or other medications that directly influence HPA axis function
* Subjects with certain lifestyle habits (i.e. working night shift) that could affect the function of the HPA axis
* History of substance dependence in the past year or meets criteria for a substance abuse disorder in the past three months.
* Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment
* Unstable or inadequately treated medical illness (e.g. diabetes, angina pectoris, hypertension) as judged by the investigator
* Participation in another drug trial within 4 weeks prior to enrollment into this study
* An absolute neutrophil count (ANC) of 1.5 x 109 per liter
* Patients who have initiated a new psychotherapy or behavioral therapy from a mental health professional in the past 3 months
* A lifetime DSM-IV history of a psychotic disorder, a bipolar disorder, or dementia.
* History of psychosurgery
* Axis II disorder
* History of seizures, excluding febrile seizures in childhood.
* Clinically relevant abnormal laboratory results.
* Patients who have received monoamine oxidase inhibitors, tricyclics, SSRIs, antipsychotics, or lithium within two weeks prior to randomization, or fluoxetine within four weeks prior to randomization.
* Electroconvulsive therapy (ECT) within three months of start of study
* History of mental retardation.
* History of major neurological illness, including any history of significant head trauma.
* Contraindications to magnetic resonance imaging, including claustrophobia and/or the presence of ferrous material that might make an MRI scan hazardous.
* Patients will be excluded from the study if they indicate at screening that they know someone who has previously participated in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
quetiapine XR treatment will be effective and safe for patients with major depression with melancholic features | 8 weeks
  Patients with major depression (N=20) will be recruited for the 8-week clinical trial of quetiapine XR 100 - 300 mg (flexible dosing). Patients who consent to participate will be referred for an initial fMRI scanning session prior to the initiation of quetiapine XR. Baseline fMRI will be obtained during the index assessment prior to initiating quetiapine XR therapy and then will be re-acquired at the final study visit at 8 weeks (the time of scheduled visits).

SECONDARY OUTCOMES:
normalization of limbic areas associated with increased salivary cortisol response to a stressful task | 8 Weeks
  successful treatment with quetiapine XR will be associated with normalization of limbic areas associated with increased salivary cortisol response to a stressful task as well as normalization on the emotional faces task differences in the melancholic group compared with healthy volunteers.
successful treatment with quetiapine XR will be associated with normalization of the salivary cortisol response to the stressful math task | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Erik Nelson, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States